CLINICAL TRIAL: NCT03996954
Title: Validation of a Smartphone-based Recorder for Detection of Cardiac Arrhythmias
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Blackpool Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Dr. Khalid Abozguia, Consultant Cardiologist and Electrophysiologist, Blackpool Teaching Hospitals NHS Foundation Trust
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: IRAS Project ID:245687
Record Dates: First submitted 2019-05-28; First posted 2019-06-25 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Cardiac Arrhythmia
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Intervention Model Description: Recordings with Alivecor and 12 lead ECGs with be acquired from patients with known arrhythmias/normal heart rhythm and blinded physicians will report on recordings and ECGs. Reports for each patient will be compared at the end of the study in order to assess diagnostic accuracy of the Alivecor to detect and differentiate between different kinds of abnormal heart rhythms.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Normal ECGs (Active Comparator): Patients with normal ECGs
  Interventions: Device: Alivecor recording
- Abnormal ECGs (Active Comparator): Patients with different kinds of abnormal heart rhythms will be enrolled in order to compare whether Alivecor can accurately differentiate between these abnormal heart rhythms and normal sinus rhythm/sinus tachycardia. Also, Alivecor diagnostic accuracy in differentiating between different kinds of arrhythmias will be assessed.
  Interventions: Device: Alivecor recording

INTERVENTIONS:
Device: Alivecor recording — Alivecor recording and ECG recording from the same patient in very close temporal proximity

SUMMARY:
The investigators will evaluate the diagnostic yield of the new AliveCor device versus a 12 lead ECG when used simultaneously to detect cardiac arrhythmia

DETAILED DESCRIPTION:
The investigators are planning to record 250 pre-defined abnormal ECGs (50 each of atrial fibrillation, atrial flutter, pre-excitation, ventricular tachycardia, , supraventricular tachycardia) and 150 control ECGs (100 sinus rhythm, 50 sinus tachycardia) using both the AliveCor Smartphone device and a 12-lead ECG. All 400 ECGs will then be read by 3 blinded reporters - a Consultant Electrophysiologist, a Consultant General Cardiologist and a General Practitioner. The output of the AliveCor automatic detection algorithm will also be recorded as a fourth reporter. The screening characteristics of all 4 reporters using the AliveCor device vs the definitive 12 lead ECG will be analysed and compared.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients >18 years
* 12 lead ECG finding of arrhythmia, manifest pre-excitation, pacing rhythm (in the EP lab), sinus rhythm or sinus tachycardia

Exclusion Criteria:

* Age <18 years
* Patients unable to or unwilling to use the device
* Patients with cardiac pacemaker, ICDs, or other implanted electronic devices

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2018-10-08 (Actual); Primary Completion 2020-10-07 (Estimated); Study Completion 2020-10-07 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of alivecor recording | Diagnostic accuracy of Alivecor recording at the end of the study which will be 2 years after study start date.
  For each patient two diagnoses of their underlying heart rhythm will be provided by blinded reporters. The percentage match of these diagnoses (the ratio of identical diagnoses to mismatch in diagnoses between ECG report and Alivecor report will be used as a measure of accuracy of the Alivecor to differentiate between different heart rhythms, using the 12 lead ECG as the gold standard for cardiac rhythm diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Khalid Abozguia, Ph.D., Principal Investigator — Blackpool Teaching Hospitals NHS Foundation Trust
Locations (1):
- Blackpool Teaching Hospitals NHS Foundation Trust, Blackpool, Lancashire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-27): https://cdn.clinicaltrials.gov/large-docs/54/NCT03996954/Prot_SAP_000.pdf